CLINICAL TRIAL: NCT05362760
Title: Combination of Abemaciclib and Endocrine Therapy in Hormone Receptor Positive HER2 Negative Locally Advanced or Metastatic Breast Cancer With Focus on Digital Side Effect Management. The MINERVA Trial - A Phase IV Trial
Brief Title: Combination of Abemaciclib and Endocrine Therapy in Hormone Receptor Positive HER2 Negative Locally Advanced or Metastatic Breast Cancer With Focus on Digital Side Effect Management
Acronym: MINERVA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, Director of the Department of Obstetrics and Gynecology, University of Ulm
Organization: University of Ulm (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MINERVA; 2021-000287-30 (EudraCT Number)
Record Dates: First submitted 2022-04-05; First posted 2022-05-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Hormone Receptor-positive Metastatic Breast Cancer; HER2-negative Metastatic Breast Cancer
Keywords: hormone receptor-positive; HER2-negative; locally advanced/metastatic breast cancer; abemaciclib; endocrine therapy; phase IV
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Aromatase Inhibitors; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Non-randomized phase 4 clinical trial with two arms (cohorts), i.e. abemaciclib plus aromatase inhibitor or abemaciclib plus fulvestrant, with patient assignment to the arms by physician's choice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Abemaciclib + Aromatase-Inhibitor (Experimental): The patients will receive Abemaciclib in combination with an Aromatase-Inhibitor (either Anastrozole, Letrozole or exemestane)
  Interventions: Drug: Abemaciclib + Aromatase Inhibitor
- Abemaciclib + Fulvestrant (Experimental): The patients will receive Abemaciclib in combination Fulvestrant
  Interventions: Drug: Abemaciclib + Fulvestrant

INTERVENTIONS:
Drug: Abemaciclib + Aromatase Inhibitor — Abemaciclib 150 mg orally every 12 hours plus Aromatase Inhibitor ( Anastrozole 1 mg, Letrozole 2.5 mg or exemestane 25 mg orally every 24 hours on Days 1 to 28 of a 28-day cycle)
  Other Names: Verzenios
  Arms: Abemaciclib + Aromatase-Inhibitor
Drug: Abemaciclib + Fulvestrant — Abemaciclib 150 mg orally every 12 hours plus Fulvestrant (500 mg intramuscularly on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond on Day 1 of a 28-day cycle)
  Other Names: Verzenios
  Arms: Abemaciclib + Fulvestrant

SUMMARY:
The MINERVA Trial aims to evaluate safety, efficacy and quality of life (QoL) for the combination of Abemaciclib with an Aromatase Inhibitor or Fulvestrant in pre- and postmenopausal patients with metastatic hormone receptor positive HER2 negative breast cancer in the first line setting.

Side effect monitoring and patient reported outcomes will be captured using the web- and app-based CANKADO digital health application. Via this user-friendly tool the patients can document their therapy side effects (e.g. diarrhea) and outcomes on a day-to-day basis. The capturing of side effects using the digital health application will be done additionally to the regular AE documentation.

Furthermore, translational research objectives of this trial include the investigation of biomarkers (ct-DNA, germline DNA) to evaluate whether they can give insights into the reasons for response, intrinsic or acquired resistance to the combined endocrine

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the trial only if they meet all the following criteria:

1. Have given written informed consent prior to any trial-specific procedures
2. Are reliable, willing to be available for the duration of the trial and are willing to follow trial procedures
3. Are female and aged ≥ 18 years
4. Diagnosis of hormone receptor positive (HR+), HER2- breast cancer. Although not required as a protocol procedure, metastatic disease should be considered for biopsy whenever possible to reassess HR and HER2 status if clinically indicated.
5. To fulfill the requirement for HR+ disease, a breast cancer must express, by immunohistochemistry (IHC), at least one of the hormone receptors (estrogen receptor [ER], progesterone receptor [PgR]) as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).
6. To fulfill the requirement of HER2- disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 by either IHC or in-situ hybridization (ISH) as defined in the relevant ASCO/CAP guidelines (Wolff et al. 2013).
7. Have locally advanced recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease
8. Indication for endocrine based therapy in the metastatic setting
9. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale
10. If central nervous system (CNS) metastases are known these have to be stable (radiotherapy finished for more than 14 days ago, no required steroid medication with more than 4 mg Dexamethasone per day)
11. Pre- and postmenopausal patients are allowed. Postmenopausal is defined as no menses for 12 months without an alternative medical cause. Women of Childbearing Potential (WOCBP, defined as not postmenopausal and not surgically or congenitally sterile) whose male partners are potentially fertile (e.g. no vasectomy) must use highly effective contraception methods for the duration of the trial and for at least 3 weeks after last dose of drugs used in the trial.Women of childbearing potential must use highly effective contraception methods for two years after the last dose of fulvestrant. Highly effective birth control methods that results in a failure rate of less than 1% per year include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner. Sexual abstinence is only considered a highly effective method if defined as refraining from heterosexual intercourse in the defined period. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the patient.
12. No prior therapy for metastatic disease (except for first line endocrine therapy for maximal 3 months prior to start of abemaciclib therapy and if no progress occurred before study entry)
13. Previous adjuvant endocrine therapy and (neo)adjuvant chemotherapy is allowed
14. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or ≤ Grade 2 peripheral neuropathy prior to registration. A washout period of at least 21 days is required between last chemotherapy dose and registration (provided the patient did not receive radiotherapy).
15. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and registration.
16. One of the following as defined by the RECIST v1. 1 (see Attachment 15.5):

    1. Measurable disease. At least one measurable lesion assessable using standard techniques by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1). Tumor evaluation according to RECIST version 1.1 (based on local assessment) has to be performed within 28 days before trial registration.
    2. Nonmeasurable bone-only disease (must be evaluable, but not necessarily measurable by RECIST). Nonmeasurable bone-only disease may include any of the following: blastic bone lesion, lytic bone lesions without a measurable soft tissue component, or mixed lytic-blastic bone lesions without a measurable soft tissue component.
17. The patient has adequate bone marrow and organ function evidenced by the following laboratory results: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, Platelet count ≥ 100 × 109/L, Hemoglobin ≥ 8 g/dL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 × ULN (≤ 3 x ULN in case of liver metastases), Total Bilirubin ≤ 1.5 × ULN (with Gilbert's syndrome max. 2 x ULN), Serum Creatinine ≤ 2.0 mg/dl or 177µmol/L, Coagulation: International Normalized Ratio (INR) ≤ 1,5
18. The patient is able to swallow oral medications
19. Willingness to use the provided CANKADO digital health application to report side effects and patient reported outcomes (The use of the CANKADO app is not mandatory for study participation, but is strongly recommended)
20. Negative pregnancy test before trial registration for women of child-bearing potential and highly effective contraception if the risk of conception exists and a negative serum pregnancy test within 7 days after the first dose of trial treatment. Pregnancy tests should be performed in premenopausal patients according to local standard

Exclusion Criteria:

Patients will be included in the trial only if they meet none of the following criteria:

1. Visceral crisis or life expectancy < 6 months
2. History of hypersensitivity reactions attributed to Abemaciclib or to other components of drug formulation
3. Prior treatment with chemotherapy in the metastatic setting or endocrine therapy in the metastatic setting (except for first line endocrine therapy in metastatic or locally advanced disease for maximal 3 months prior to start of abemaciclib therapy and if no progress occurred before study entry)
4. Patient not eligible for endocrine based therapy
5. Any concurrent severe, uncontrolled systemic disease, social or psychiatric condition that might interfere with the planned treatment and with the patient's adherence to the protocol
6. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this trial (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
7. Prior treatment with a CDK4/6 inhibitor for metastatic or locally advanced disease (first-line treatment with a CDK 4/6 inhibitor (Ribociclib/Palbociclib) in the metastatic setting is allowed only if terminated due to toxicity after max 3 months and no progression occurred before study entry. Prior treatment with a CDK 4/6 inhibitor in the neo-/adjuvant setting is allowed.)
8. 8. Treatment with any other investigational agents within four weeks or 5 half-lives prior to trial registration, whichever is longer
9. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
10. Females who are pregnant or lactating
11. Legal incapacity or limited legal capacity
12. History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years.
13. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating trial treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
14. Prior systemic anti-cancer therapy within the last 21 days prior to start of trial treatment except for first-line endocrine therapy in metastatic or locally advanced disease (see above)
15. Radiotherapy within the last 14 days prior to registration
16. Patient has had major surgery within 14 days prior to trial registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Time from date of trial registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  PFS, defined as the time from date of trial registration until progressive disease (PD) or death from any cause, whichever comes first (as defined by RECIST guideline version 1.1). If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.

SECONDARY OUTCOMES:
Adverse Events | From obtaining informed consent until progressive disease (PD) or up to 30 days after end of trial treatment
  Adverse Events assessed by investigator (type, frequency, severity (graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0)), seriousness)
Patient-reported side effects | From first dose of study medication up to 30 days after end of trial treatment
  Additional capture of Patient-Reported side effects on a daily basis via CANKADO PRO-React (patient diary).
Patient-reported global health status | From first dose of study medication up to 30 days after end of trial treatment
  Daily self-assessment of global health status using the visual analogue scale (EQ-VAS, based on the EQ-5D questionnaire) via CANKADO. The EQ-VAS scale ranges from 0 (the worst possible health status to 100 (the best possible health status).
Frequency of hospitalizations | Time from date of registration for the trial through study completion (4 years after date of First Patient In)
  Frequency of hospitalizations during study treatment
Patient reported European Organisation for Research and Treatment of Cancer Quality of Life C30 questionaire (EORTC QLQ-C30) | At baseline, at 3, 6, 9, 12, 18, 24 months
  Patient reported quality of life as assessed with the EORTC QLQ-C30 questionnaire. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Patient reported European Organisation for Research and Treatment of Cancer Quality of Life B23 breast cancer module questionaire (EORTC QLQ-BR23) | At baseline, at 3, 6, 9, 12, 18, 24 months
  Patient reported quality of life as assessed with the EORTC QLQ-BR23 questionnaire. The QLQ-B23 breast cancer module incorporates five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Clinical benefit rate (CBR) | Time from date of registration for the trial until 24 weeks of study treatment
  CBR defined as percentage of patients with complete response, partial response or stable disease
Overall Survival (OS) | Time from date of trial registration until date of death due to any cause, assessed up to 48 months
  Overall survival (OS) defined as the time from date of trial registration until date of death due to any cause. If a patient is not known to have died, survival is censored at the date of last contact.
Objective Response Rate (ORR) | Time from date of registration for the trial through study completion (4 years after date of First Patient In)
  ORR defined as percentage of patients with complete or partial response as defined by RECIST 1.1
Number of patients with primary progression | Time from date of registration for the trial until first imaging after 12 weeks
  Number of patients with primary progression, defined as number of patients with disease recurrence within 12 weeks after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Rack, Prof. Dr., Principal Investigator — Department of Gynecology and Obstetrics, University Hospital Ulm, Germany
Locations (54):
- Germany (52):
  - Kliniken Ostalb gkAöR, Aalen
  - Klinikum St. Marien Kommunalunternehmen - AöR Der Stadt Amberg, Amberg
  - Klinikum Aschaffenburg-Alzenau gGmbH, Aschaffenburg
  - Gemeinschaftspraxis Dr. Heinrich / Dr. Bangerter, Augsburg
  - Universitätsklinikum Augsburg A.d.ö.R, Augsburg
  - MediOnko-Institut GbR, Berlin
  - Hämatologikum Biberach, Biberach
  - Gynäkologisches Zentrum Bonn - Friedensplatz, Bonn
  - Studien GbR Braunschweig, Braunschweig
  - Hämato-Onkologische Praxis im Medicum, Bremen
  - St. Elisabeth-Krankenhaus GmbH, Cologne
  - Onkologisches Zentrum Donauwörth, Donauwörth
  - Gemeinschaftspraxis, Dresden
  - Onkozentrum Dresden, Dresden
  - MVZ Medical Center Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Internistische Praxis Ehingen, Ehingen
  - Universitätsklinikum Erlangen, Erlangen
  - St. Antonius-Hospital, Eschweiler
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Krankenhäuser Landkreis Freudenstadt gGmbH, Freudenstadt
  - Internistische Gemeinschaftspraxis, Friedrichshafen
  - Klinikum Garmisch-Partenkirchen GmbH, Garmisch-Partenkirchen
  - Main-Kinzig-Kliniken gGmbH Gelnhausen, Gelnhausen
  - Gemeinschaftspraxis und Tagesklinik Halle, Halle
  - Albertinen-Krankenhaus, Hamburg
  - Sana Klinikum Hameln-Pyrmont, Hamelin
  - Frauenärzte am Bahnhofsplatz, Hildesheim
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel GmbH, Kassel
  - Klinikverbund Kempten-Oberallgäu gGmbH, Kempten
  - Klinikum Konstanz, Konstanz
  - ZAGO- Zentrum für ambulante gynäkologische Onkologie, Krefeld
  - Krankenhausgesellschaft St. Vincenz mbH, Limburg
  - Praxis für gynäkologische Onkologie / Prof. Dr. med. Ulrike Nitz / Raquel von Schumann, Mönchengladbach
  - Kliniken Ostalb gkAöR, Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - LMU - Klinikum der Universität München, München
  - München Klinik gGmbH Harlaching, München
  - TZN-Tumorzentrum Niederrhein GmbH, Neuss
  - Klinikum Nürnberg Nord, Nuremberg
  - medius KLINIK NÜRTINGEN, Nürtingen
  - Praxis Dr. Guth, Plauen
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Klinikum Rheine, Rheine
  - GPR Gesundheits- und Pflegezentrum Rüsselsheim gGmbH, Rüsselsheim am Main
  - Diakoneo Diak-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Clinical Research Stolberg GmbH, Stolberg
  - Gynäkologie Kompetenzzentrum Stralsund, Stralsund
  - Universitätsfrauenklinik Tübingen, Tübingen
  - University Hospital Ulm Gynecology/Obstetrics, Ulm
  - St. Josefs-Hospital, Wiesbaden
- Switzerland (2):
  - Spital Wallis, Brig
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No